CLINICAL TRIAL: NCT05905458
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-designed Phase II Study to Evaluate the Efficacy and Safety of HRS9950 Tablets in Chronic Hepatitis B Patients Who Are Virologically Suppressed on Nucleoside or Nucleotide Analogues (NAs)
Brief Title: A Phase II Clinical Study of the Efficacy and Safety of HRS9950 Tablets in Chronic Hepatitis B Patients Who Are Virologically Suppressed on Nucleoside or Nucleotide Analogues (NAs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9950-201
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: HRS9950 tablets (Low dose) (Experimental)
  Interventions: Drug: HRS9950 tablets
- Treatment group B: HRS9950 tablets (High dose) (Experimental)
  Interventions: Drug: HRS9950 tablets
- Placebo Comparator: Treatment group C (Placebo Comparator)
  Interventions: Drug: HRS9950 placebo tablets

INTERVENTIONS:
Drug: HRS9950 tablets — HRS9950 tablets, oral, once a week, low dose
  Arms: Treatment group A: HRS9950 tablets (Low dose)
Drug: HRS9950 tablets — HRS9950 tablets, oral, once a week, high dose
  Arms: Treatment group B: HRS9950 tablets (High dose)
Drug: HRS9950 placebo tablets — HRS9950 placebo tablets, oral, once a week.
  Arms: Placebo Comparator: Treatment group C

SUMMARY:
To evaluate the efficacy and safety of HRS9950 tablets in chronic hepatitis B patients who are virologically suppressed on nucleoside or nucleotide analogues (NAs).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the body mass index standard among 18.0 to 30 kg/m2;；
2. Chronic hepatitis B defined as HBV infection documented for at least 6 months prior to screening;
3. Virologically suppressed on nucleoside or nucleotide analogues treatment with HBV DNA below the lower limit of quantitation;
4. On commercially available NAs monotherapy for at least 24 weeks before randomization, and the dosing regimen remained unchanged for at least 12 weeks before randomization;
5. Need to take effective contraceptive measures；
6. Volunteer to sign an informed consent.

Exclusion Criteria:

1. History of cirrhosis or clinical evidence of hepatic decompensation, confirmed or suspected liver cancer, with other liver diseases other than chronic hepatitis B that may affect the evaluation of the study;
2. With autoimmune disease;
3. With poorly-controlled diabetes, thyroid disease requiring clinical intervention, clinically significant thyroid dysfunction, neurological or psychiatric disorder, severe lung disease, chronic renal disease or retinopathy;
4. History of solid organ transplantation or hematopoietic stem cell transplantation;
5. Poorly-controlled hypertension, clinically significant and unstable or uncontrolled severe cardiovascular and cerebrovascular diseases;
6. Malignant tumors were diagnosed within 5 years prior to randomization；
7. Infection requiring intervention within 4 weeks prior to randomization;
8. Major trauma or major surgery within the 12 weeks prior to randomization, or surgical plans or other treatment during the study period which the investigators determined may influence the evaluation of the study results;
9. Laboratory tests during the screening period were obviously abnormal;
10. Prolonged ECG QTc interval (male > 450ms, female > 470ms) or other clinically significant abnormal results that may pose significant safety risks to subjects during the screening period;
11. History of drug use, alcohol or drug abuse in the 12 months prior to randomization;
12. Participated in clinical study of other drugs (received experimental drugs);
13. Pregnant or nursing women;
14. Allergic to a drug ingredient or component;
15. Other reasons for ineligibility as judged by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Change in mean log10 serum hepatitis B surface antigen levels from baseline to week 24 | Week 24

SECONDARY OUTCOMES:
Changes from baseline in mean log10 serum hepatitis B surface antigen levels | Pre-specified time points up to 48 weeks
Proportion of subjects with at least one log10 decline from baseline in serum hepatitis B surface antigen | Pre-specified time points up to 48 weeks
Proportion of subjects with serum hepatitis B surface antigen loss | Pre-specified time points up to 48 weeks
Proportion of subjects with serum hepatitis B surface antigen seroconversion | Pre-specified time points up to 48 weeks
Proportion of subjects with hepatitis B e-antigen loss | Pre-specified time points up to 48 weeks
Proportion of subjects with serum hepatitis B e-antigen seroconversion | Pre-specified time points up to 48 weeks
Proportion of subjects with virologic breakthrough | Pre-specified time points up to 48 weeks
Proportion of subjects with drug resistance | Pre-specified time points up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided